CLINICAL TRIAL: NCT03809013
Title: A Open-label, Single-arm, Multicenter, Phase II Study of RC48-ADC to Evaluate the Efficacy and Safety of Subjects With HER2 Overexpressing Locally Advanced or Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C009
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC (Experimental): Participants will be treated with RC48-ADC 2.0 mg/kg, once every 2 weeks (Q2W) until investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or participant's decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC

INTERVENTIONS:
Drug: RC48-ADC — 2.0mg/kg IV every 2 weeks
  Other Names: Recombinant Humanized anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection

SUMMARY:
This study will evaluate the efficacy and safety of intravenous RC48-ADC in patients with HER2 overexpressing locally advanced or metastatic urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years.
* Predicted survival ≥ 12 weeks.
* Diagnosed with histologically or cytologically-confirmed locally advanced or metastatic urothelial cancer, originate from bladder, renal pelvis, ureter and urinary tract.
* Unresectable or disease progression (i.e. locally advanced/metastasis) after surgery and at least regular chemotherapy including gemcitabine,cisplatin AND paclitaxel. Disease progression within 6 months of the completion of neo-adjuvant and adjuvant chemotherapy with gemcitabine, cisplatin AND paclitaxel is also eligible.
* Measurable lesion according to RECIST 1.1.
* HER2 overexpressing (i.e. IHC 2+ or 3+) as confirmed by the central lab. Primary or metastatic tumor sample will be provided for HER2 test.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function, evidenced by the following laboratory results within 7 days prior to the study treatment:

Cardiac ejection fraction ≥ 50 %. Hemoglobin ≥ 9g/dL; Absolute neutrophil count ≥ 1.5×109 /L Platelets ≥ 100×109 /L; Total bilirubin ≤ 1.5× ULN; AST and ALT ≤ 2.5×ULN and ≤ 5 × ULN with hepatic metastasis; Serum creatinine ≤1.5×ULN.

* All female subjects will be considered to be of child-bearing potential unless they are postmenopausal, or have been sterilized surgically.Female subjects of child-bearing potential must agree to use two forms of highly effective contraception. Male subjects and their female partner who are of child-bearing potential must agree to use two forms of highly effective contraception.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Known hypersensitivity to the components of Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate.
* Toxicity of previous anti-tumor treatment not recovered to CTCAE Grade 0-1 (with exception of Grade 2 alopecia).
* Pleural or abdominal effusion with clinical symptoms that requires ongoing treatment.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* Currently known active infection with HIV or tuberculosis.
* Diagnosed with HBsAg, HBcAb positive and HBV DNA copy positive, or HCVAb positive.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* known central nervous system metastases.
* Uncontrolled hypertension, diabetes, Interstitial lung Disease, or COPD;
* Treated with systemic treatment (e.g. immunomodulators, corticosteroids or immunosuppressants) for the autoimmune disease within 2 years prior to the study treatment.
* NYHA Class III heart failure.
* Pregnancy or lactation.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate （ORR）as assessed by the Independent Review Committee | 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Objective Response Rate（ORR）as assessed by investigator | 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Progression Free Survival (PFS) | 24 months
  PFS was defined as the time from the first administration of study treatment to the first occurrence of disease progression as determined by investigator using RECIST v1.1 or death from any cause, whichever comes first
Duration of Objective Response (DOR) | 24 months
  DOR was defined as the time from first documented OR to first documented PD or death from any cause, whichever occurred earlier
Disease control rate (DCR) | 24 months
  DCR was defined as the percentage of participants with a complete response (CR), partial response (PR), or stable disease (SD)
Overall survival (OS) | 24 months
  OS was defined as the time from the first administration of study treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Ph.D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (8):
- China (8):
  - Anhui Cancer Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sheng X, Wang L, He Z, Shi Y, Luo H, Han W, Yao X, Shi B, Liu J, Hu C, Liu Z, Guo H, Yu G, Ji Z, Ying J, Ling Y, Yu S, Hu Y, Guo J, Fang J, Zhou A, Guo J. Efficacy and Safety of Disitamab Vedotin in Patients With Human Epidermal Growth Factor Receptor 2-Positive Locally Advanced or Metastatic Urothelial Carcinoma: A Combined Analysis of Two Phase II Clinical Trials. J Clin Oncol. 2024 Apr 20;42(12):1391-1402. doi: 10.1200/JCO.22.02912. Epub 2023 Nov 21. PMID 37988648